CLINICAL TRIAL: NCT05506852
Title: Training Executive Control in Cognitively Healthy Aging: the Web-based Breakfast Game
Brief Title: Using Teleneuropsychology to Optimize Cognition in Healthy Aging: the Web-based Breakfast Game
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sharon Sanz Simon, Principal Investigator, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAT4773; 1K99AG078561-01 (NIH)
Record Dates: First submitted 2022-07-25; First posted 2022-08-18 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Healthy Aging
Keywords: cognition; cognitive training; non-pharmacological intervention; video game; cognitive enhancement; computer-based; teleneuropsychology; computerized; attention control; executive control; cognitive decline; multi-tasking
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be aware of the difference across the two conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strategy Training (Experimental): Participants will play the Breakfast Game with training strategy.
  Interventions: Behavioral: Web-based training strategy
- Regular Approach (Active Comparator): Participants will play the Breakfast Game without training strategy.
  Interventions: Behavioral: Web-based regular training (no strategy)

INTERVENTIONS:
Behavioral: Web-based training strategy — Participants will undergo a web-based training protocol where they will play an online game that simulates a breakfast environment and will perform everyday activities as "cooking" and "setting tables" in a multi-tasking fashion. Participants will learn to play the game using specific strategies, in order to optimize the performance.
  Other Names: Experimental intervention
  Arms: Strategy Training
Behavioral: Web-based regular training (no strategy) — Participants will undergo a web-based training protocol where they will play an online game that simulates a breakfast environment and will perform everyday activities as "cooking" and "setting tables" in a multi-tasking fashion. Participants will learn to play the game under regular game instructions.
  Other Names: Control intervention
  Arms: Regular Approach

SUMMARY:
Executive control processes involve initiate, coordinate, synchronize, and regulate elemental cognitive functions for the conduct of goal-directed behavior. The proposed research investigates whether exposure to a web-based training protocol designed to enhance executive control processes will improve cognitive performance in cognitively healthy older adults.

DETAILED DESCRIPTION:
The proposed research investigates whether exposure to a web-based training protocol designed to enhance executive control / multi-tasking abilities will improve cognitive performance in healthy older adults. Cognitively normal adults aged 60-75 will be randomized into two experimental groups: 1) Web-based game with training strategy; 2) Web-based game without training strategy (Active Control). All participants (groups 1 and 2) will be instructed to play the complex, high-demand online game, Breakfast Game, for 14 one-hour sessions over 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-75
* Willingness to adhere to training protocol
* Adequate English proficiency

Exclusion Criteria:

* Low test scores (below 26 on the Montreal Cognitive Assessment)
* Known history of cognitive impairment, dementia, stroke, seizure disorder, or other neuropsychiatric condition judged to impact cognitive performance.
* Taking medications known to influence cognitive performance.
* Sensory (e.g. visual, auditory) or physical (e.g. severe arthritic, orthopedic, neurologic) impairment incompatible with use of a standard computer workstation.
* Enrolled in a concurrent study that could affect the outcome of this study.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in the Breakfast Game performance: Number of Tables Set Score | Training session 2, week 2; training 13, approximately 6 weeks.
  Change in the total number of tables set. In the computerized task, participants are asked to set tables for four guests, when finished, one point is given. Higher scores represent a better outcome.
Changes in the Breakfast Game performance: Cooking time Range of Stop Times scores. | Training session 2, week 2; training 13, approximately 6 weeks.
  Change in cooking time (milliseconds) between food items. In the computerized task, participants are asked to cook different food types. Scores reflect is the difference between the first and last food item stopped cooking. Lowers scores (closest to zero) represent a better outcome.
Change in Breakfast Game performance: Cooking Time Discrepancy scores | Training session 2, week 2; training 13, approximately 6 weeks.
  Change in cooking time (milliseconds) in each food type. In the computerized task, participants are asked to cook different food types. Scores reflect the average absolute values of the difference between the required and actual cooking time of each item. Lowers scores (closest to zero) represent a better outcome.
Transfer to complex executive/attention control measure (Proximal outcome). | Within the 2 weeks before intervention starts; and 6th week, after the last (13th) training session.
  Accuracy on Alphanumeric Task

SECONDARY OUTCOMES:
Transfer to executive functions composite measure (Distal outcome) | Within the 2 weeks before intervention starts; and 6th week, after the last (13th) training session.
  Average z-score computed with tests involving working memory, inhibitory control, cognitive flexibility (Letter-Number, Wisconsin, and Stroop)
Transfer to divided attention / speed measure (Distal outcome) | Within the 2 weeks before intervention starts; and 6th week, after the last (13th) training session.
  Accuracy and reaction time on the Useful Field of View.
Transfer to episodic memory/learning measure (Distal outcome) | Within the 2 weeks before intervention starts; and 6th week, after the last (13th) training session.
  Accuracy and reaction time on list learning test.
Transfer to the General Self-efficacy Scale (Distal outcome) | Within the 2 weeks before intervention starts; and 6th week, after the last (13th) training session.
  Scores on a scale that measures perception about self-efficacy. Total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Transfer to Beck Depression Inventory (Distal outcome) | Within the 2 weeks before intervention starts; and 6th week, after the last (13th) training session.
  Score on a scale that measures depression symptoms. Total score ranges between 0 and 63, with a higher score indicating more depression symptoms.
Transfer to Beck Anxiety Inventory (Distal outcome) | Within the 2 weeks before intervention starts; and 6th week, after the last (13th) training session.
  Score on a scale that measures anxiety symptoms. Total score ranges between 0 and 63, with a higher score indicating more anxiety symptoms.
Transfer to Cognitive Failure Questionnaire (Distal outcome) | Within the 2 weeks before intervention starts; and 6th week, after the last (13th) training session.
  Score on a scale reflecting frequency/difficulties on complex daily life activities. Total score ranges between 0 and 100, with a higher score indicating more cognitive difficulties in every daylife.
Transfer to Cognition-Leisure Questionnaire (Distal outcome) | Within the 2 weeks before intervention starts; and 6th week, after the last (13th) training session.
  Score on a scale reflecting engagement/frequency in leisure & cognitive activities.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Sanz Simon, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by the principal investigator.